CLINICAL TRIAL: NCT07259343
Title: Effect of Glycomacropeptide on Clinical Manifestations of Atopic Dermatitis in Children: a Pilot Study
Brief Title: Effect of an Emollient Cream Containing a Milk Bioactive Peptide on Clinical Signs, Pruritus and Bacterial Colonization of Mild Atopic Dermatitis Skin Lesions in Pediatric Population
Acronym: AD-GMP-SCORAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Aguascalientes (Other)
Responsible Party: Principal Investigator, Eva María Salinas Miralles, Professor and Researcher, C, Universidad Autónoma de Aguascalientes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COB-UAA/09/2024; PIBB26-2 (Other Grant/Funding Number: Autonomous University of Aguascalientes)
Record Dates: First submitted 2025-09-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis (AD)
Keywords: glycomacropeptide; eczema; priritus; Staphylococcus
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — caseinomacropeptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical administration of an emollient cream formulated with glycomacropeptide (Experimental): Topical administration of an emollient cream formulated with 5% glycomacropeptide, applied twice daily for 4 weeks, restricted to affected skin areas, in pediatric patients with atopic dermatitis
  Interventions: Other: glycomacropeptide
- Topical administration of the emollient cream formulated without glycomacropeptide (Active Comparator): Topical administration of the emollient vehicle cream without glycomacropeptide, applied twice daily for 4 weeks to affected skin areas, in pediatric patients with atopic dermatitis
  Interventions: Other: emollient cream

INTERVENTIONS:
Other: glycomacropeptide — Topical application of an emollient cream formulated with 5% glycomacropeptide, applied twice daily for 4 weeks
  Arms: Topical administration of an emollient cream formulated with glycomacropeptide
Other: emollient cream — Topical administration of an emollient cream, applied twice daily for 4 weeks to affected skin areas
  Arms: Topical administration of the emollient cream formulated without glycomacropeptide

SUMMARY:
The goal of this clinical trial is to evaluate the protective effect of glycomacropeptide on the clinical signs and symptoms of atopic dermatitis in children aged 2 to 12 years, and to determine if topical administration of glycomacropeptide is associated with a lower colonization by Staphylococcus species on the skin. The main questions that it aims to answer are:

* Does glycomacropeptide reduce the signs and symptoms related to atopic dermatitis in the pediatric population?
* Does glycomacropeptide modify the colonization of Staphylococcus species in atopic dermatitis lesions in the pediatric population? Researchers will compare an emollient cream containing glycomacropeptide with an emollient cream without glycomacropeptide to evaluate whether treatment with glycomacropeptide achieves a greater reduction in the clinical severity and pruritus of atopic dermatitis and a lower bacterial colonization compared with the exclusive use of emollients.

Participants will:

* Read and sign the informed consent
* Undergo a prick test at the first visit to ensure no reaction to the treatment components
* Receive the assigned treatment (glycomacropeptide cream or emollient cream), which must be applied twice daily only to atopic dermatitis lesions.
* Visit the clinic once a week for 4 weeks for follow-up and SCORAD assessments, and for skin sample collection by stripping at first and last visit.

DETAILED DESCRIPTION:
Atopic dermatitis is a chronic and recurrent skin disease characterized by intense pruritus, dry skin, inflammation, and, in some cases, eczema. Although it can occur at any age, it is more common in childhood, with a global prevalence estimated between 5% and 20% in children, and approximately 7.3% in adults. Its impact on quality-of-life ranges from mild discomfort to significant sleep disturbances and limitations in daily activities.

The pathogenesis of atopic dermatitis is associated with structural and functional impairment of the epidermis, leading to inflammation, dysregulation of T helper cells (Th1/Th2), increased immunoglobulin E production, and mast cell hyperactivity, all of which exacerbate barrier abnormalities. The most common barrier defect is decreased production of filaggrin or other stratum corneum proteins, contributing to xerosis and increased susceptibility to infections. In addition, reduced production of antimicrobial peptides facilitates bacterial colonization.

Current treatment of atopic dermatitis relies on emollients, topical corticosteroids, and topical or systemic calcineurin inhibitors, depending on disease severity and persistence. However, prolonged use of these drugs can result in adverse effects such as burning, hypertrichosis, telangiectasias, skin atrophy, acne, folliculitis, contact dermatitis, nephrotoxicity, hepatotoxicity, seizures, and neoplasms. Therefore, there is a need for alternative treatments that can reduce quantity and time for drugs and promote patient recovery.

Glycomacropeptide is a 64-amino acid peptide derived from bovine casein during cheese production by chymosin or during milk digestion by pepsin. It is highly glycosylated, mainly at serine and threonine residues, with tetra-saccharides containing sialic acid as a key component of its bioactivity. Clinical studies have demonstrated the safety of oral glycomacropeptide in humans, and multiple biological activities have been described, including anti-inflammatory and anti-allergic effects in preclinical models of asthma, urticaria, food allergy, and atopic dermatitis.

About skin, glycomacropeptide has shown beneficial effects on keratinocytes, protecting them against apoptosis, inflammation, and oxidative stress, while promoting their migration and proliferation, processes that support skin repair in atopic conditions. Glycomacropeptide also inhibits mast cell and macrophage activation, key immune cells abundant in atopic dermatitis lesions that contribute to chronic inflammation.

Atopic dermatitis is associated with skin dysbiosis, characterized by reduced bacterial diversity and overgrowth of Staphylococcus aureus. In vitro studies from our laboratory demonstrate that glycomacropeptide does not promote the growth of S. aureus or Staphylococcus epidermidis. Instead, it inhibits S. aureus adhesion to human keratinocytes and, in contrast, enhances S. epidermidis adhesion, a commensal species that contributes to skin homeostasis. Furthermore, glycomacropeptide reduces the ability of S. aureus to form biofilms, a key persistence mechanism.

These findings support the potential of glycomacropeptide as a topical therapeutic candidate for atopic dermatitis, acting through modulation of inflammation, skin repair, and modulation of the microbiota.

This is a randomized, parallel, double-blind clinical trial. The primary objective is to evaluate the protective effect of topical glycomacropeptide on the clinical signs and symptoms of atopic dermatitis in children.

The secondary objectives are:

1. To determine whether topical glycomacropeptide is safe and well tolerated in children with atopic dermatitis.
2. To determine whether topical glycomacropeptide is associated with changes in the severity of atopic dermatitis lesions and the extent of eczema, based on the SCORAD index.
3. To determine whether topical glycomacropeptide decreases pruritus associated with eczema and improves sleep duration.
4. To determine whether topical glycomacropeptide is associated with reduced S. aureus colonization on the skin.

The main questions this study aims to answer are:

* Does glycomacropeptide reduce the signs and symptoms related to atopic dermatitis in the pediatric population?
* Does glycomacropeptide modify the colonization of Staphylococcus species in atopic dermatitis lesions in the pediatric population? Study Population. Children aged 2 to 12 years with a diagnosis of atopic dermatitis confirmed by the Hanifin and Rajka criteria, and classified as mild according to the SCORAD index (<25 points). Participants will be excluded if they fall outside the age range, present a SCORAD score >25, have concomitant dermatoses, a history of hypersensitivity or anaphylaxis to any treatment components, inability to attend follow-up visits or adhere to the treatment schedule, or any clinical condition deemed unsuitable by the investigator.

Data verification procedures will be implemented to ensure precision and consistency. The database will include predefined rules for ranges and logical consistency checks (for example, age 2-12 years, SCORAD <25 at inclusion). Data that fall outside the expected range or are inconsistent with other fields will be flagged for review and corrected or canceled, as the case may be.

Recruitment Strategy. Enrollment will be carried out through collaboration with local pediatric, allergy and immunology, and dermatology medical associations. Additionally, screening campaigns will be conducted in primary schools to identify potential participants, followed by guardian consent discussions.

Sample Size and Interventions. A total of 20 eligible participants will be randomly assigned into two groups:

1. Emollient cream with glycomacropeptide.
2. Emollient cream without glycomacropeptide (control). Both formulations will be applied topically to atopic dermatitis lesions twice daily for 4 weeks. Participants will attend weekly follow-up visits for clinical evaluation and SCORAD assessment. At the first visit, a prick test will be performed to rule out hypersensitivity to cream components. In addition, skin samples will be obtained by stripping at baseline and at the final visit to quantify colonization by Staphylococcus species.

Data dictionary for study variables:

The independent variables of the study include:

* Sex: Defined as morphological differences between male and female. It will be obtained from the clinical record and classified as male or female.
* Age: Defined as the time period between birth and participation in the study. It will be obtained from the clinical record and expressed in complete years, with an expected range of 2 to 12 years.

The dependent variables of the study include:

* Atopic dermatitis diagnosis: Defined as the presence of a chronic and recurrent skin disease, confirmed by fulfilling at least three major and three minor Hanifin and Rajka criteria. Classified as present or absent.
* Severity of atopic dermatitis: Defined as the objective and subjective clinical characteristics of the disease, measured using the SCORAD Index. Severity will be categorized as mild (<25), moderate (25-50), or severe (>50).
* Exacerbation: Defined as the increase or recurrence of symptoms after a symptom-free period, also measured by the SCORAD Index, and classified as mild, moderate, or severe according to the same cut-off points.
* Remission period: Defined as the duration of absence of symptoms of atopic dermatitis. It will be measured in days, based on clinical evaluations.
* Exacerbation period: Defined as the duration of symptom exacerbation. It will be measured in days, based on clinical evaluations.
* Colonization by S. aureus: Defined as the presence and quantity of this opportunistic gram-positive bacterium in atopic dermatitis lesions. It will be measured through skin stripping samples analyzed by culture or PCR, expressed as copies of S. aureus femA gene per ng of total DNA.
* Ratio of S. aureus to S. epidermidis: Defined as the relationship between a pathogenic species and a commensal species of the cutaneous microbiota. It will be measured through skin stripping samples analyzed by culture or PCR, expressed as the ratio of DNA femA gene copies (S. aureus/S. epidermidis).
* Prick test: Defined as a skin test that exposes mast cells to allergens to detect sensitization. It will be recorded as positive when a wheal of ≥3 mm larger than the negative control is observed, and negative otherwise.

Data Collection. A quality assurance plan will be implemented to ensure precision and completeness of the collected data. A pediatric allergologist and the principal investigator will supervise adherence to the protocol at each participant in all clinical evaluations, and laboratory procedures will be performed according to standardized protocols.

All missing, unavailable, or uninterpretable data will be recorded as "missing." Data inconsistencies or out-of-range results will also be considered missing. The primary analysis will use the available data without imputation. Data will be analyzed using Prism GraphPad software, applying appropriate statistical methods according to the variables of interest.

All study records will be available for review by the ethics committee or external auditors if required.

Data Analysis. The statistical analysis will include descriptive statistics to summarize baseline characteristics of participants, including means, standard deviations, frequencies, and percentages, as appropriate. Comparisons between study groups will be performed using Chi-square tests. Continuous variables, including SCORAD index scores, bacterial colonization (S. aureus load and S. aureus/S. epidermidis ratio), and clinical outcomes such as duration of remission and exacerbation periods, will be compared between groups using Student's t tests. Statistical significance will be set at p < 0.05, and analyses will be conducted using Prism GraphPad software.

Final Report and Dissemination. Based on the results, a final study report will be prepared and a scientific manuscript will be drafted for potential publication.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 12 years.
* Clinical diagnosis of atopic dermatitis according to Hanifin and Rajka criteria.
* Mild atopic dermatitis with SCORAD <25 points.
* Written informed consent signed by parents or legal guardian.

Exclusion Criteria:

* Age younger than 2 years or older than 12 years.
* Moderate to severe atopic dermatitis (SCORAD >25 points).
* Presence of other dermatoses in addition to atopic dermatitis.
* Background of hypersensitivity or anaphylaxis to any components of the vehicle cream.
* Allergy or hypersensitivity to glycomacropeptide.
* Inability to attend follow-up medical consultations or to adhere to the treatment schedule.
* Any clinical reason determined by the clinical investigator that makes the child unsuitable for the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in SCORAD index | From enrollment to the end of treatment at 4 weeks
  Change in severity and extent of atopic dermatitis lesions assessed by the SCORAD (Scoring Atopic Dermatitis) index

SECONDARY OUTCOMES:
Change in pruritus intensity | From enrollment to the end of treatment at 4 weeks
  Change in pruritus intensity assessed by visual analogue scale where 0 in no itch and 10 is the worst imaginable itch
Change in sleep quality | From enrollment to the end of treatment at 4 weeks.
  Change in sleeplessness assessed by visual analogue scale where 0 in no sleeplessness and 10 is the worst imaginable sleeplessness
Change in staphylococcal skin colonization by Staphylococcus aureus and Staphylococcus epidermidis | From enrollment to the end of treatment at 4 weeks
  Difference in the amount of Staphylococcus aureus and Staphylococcus epidermidis in lesional skin samples
Safety of glycomacropeptide topical application | From enrollment to the end of treatment at 4 weeks
  Record and report of any adverse cutaneous reactions observed in patients receiving treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Salinas, PhD, Principal Investigator — Universidad Autónoma de Aguascalientes
Locations (1):
- Universidad Autónoma de Aguascalientes, Aguascalientes, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual participant data, including SCORAD scores, pruritus intensity, sleep quality, and microbiological findings
Time Frame: Data will be available after publication of primary results and for up to 5 years.
Access Criteria: Upon reasonable request from qualified researchers for academic purposes

REFERENCES:
- [Background] Ogai K, Nagase S, Mukai K, Iuchi T, Mori Y, Matsue M, Sugitani K, Sugama J, Okamoto S. A Comparison of Techniques for Collecting Skin Microbiome Samples: Swabbing Versus Tape-Stripping. Front Microbiol. 2018 Oct 2;9:2362. doi: 10.3389/fmicb.2018.02362. eCollection 2018. PMID 30333815
- [Background] Ogai K, Shibata K, Takahashi N, Ogura K, Okamoto S, Sugama J. Amplicon-based skin microbiome profiles collected by tape stripping with different adhesive film dressings: a comparative study. BMC Microbiol. 2021 Feb 18;21(1):54. doi: 10.1186/s12866-021-02122-4. PMID 33602131
- [Background] Oppenheimer J, Nelson HS. Skin testing: a survey of allergists. Ann Allergy Asthma Immunol. 2006 Jan;96(1):19-23. doi: 10.1016/S1081-1206(10)61034-4. PMID 16440527
- [Background] Nelson HS, Knoetzer J, Bucher B. Effect of distance between sites and region of the body on results of skin prick tests. J Allergy Clin Immunol. 1996 Feb;97(2):596-601. doi: 10.1016/s0091-6749(96)70304-4. PMID 8621844
- [Background] Manguy J, Shields DC. Implications of kappa-casein evolutionary diversity for the self-assembly and aggregation of casein micelles. R Soc Open Sci. 2019 Oct 16;6(10):190939. doi: 10.1098/rsos.190939. eCollection 2019 Oct. PMID 31824707
- [Background] Zhou H, Tan X, Chen G, Liu X, Feng A, Liu Z, Liu W. Extracellular Vesicles of Commensal Skin Microbiota Alleviate Cutaneous Inflammation in Atopic Dermatitis Mouse Model by Re-Establishing Skin Homeostasis. J Invest Dermatol. 2025 Feb;145(2):312-322.e9. doi: 10.1016/j.jid.2023.02.023. Epub 2023 Mar 11. PMID 36907322
- [Background] Koh LF, Ong RY, Common JE. Skin microbiome of atopic dermatitis. Allergol Int. 2022 Jan;71(1):31-39. doi: 10.1016/j.alit.2021.11.001. Epub 2021 Nov 24. PMID 34838450
- [Background] Jimenez M, Cervantes-Garcia D, Munoz YH, Garcia A, Haro LM Jr, Salinas E. Novel Mechanisms Underlying the Therapeutic Effect of Glycomacropeptide on Allergy: Change in Gut Microbiota, Upregulation of TGF-beta, and Inhibition of Mast Cells. Int Arch Allergy Immunol. 2016;171(3-4):217-226. doi: 10.1159/000453035. Epub 2017 Jan 4. PMID 28049206
- [Background] Gallegos-Alcala P, Jimenez M, Cervantes-Garcia D, Cordova-Davalos LE, Gonzalez-Curiel I, Salinas E. Glycomacropeptide Protects against Inflammation and Oxidative Stress, and Promotes Wound Healing in an Atopic Dermatitis Model of Human Keratinocytes. Foods. 2023 May 9;12(10):1932. doi: 10.3390/foods12101932. PMID 37238750
- [Background] Jimenez M, Munoz FC, Cervantes-Garcia D, Cervantes MM, Hernandez-Mercado A, Barron-Garcia B, Moreno Hernandez-Duque JL, Rodriguez-Carlos A, Rivas-Santiago B, Salinas E. Protective Effect of Glycomacropeptide on the Atopic Dermatitis-Like Dysfunctional Skin Barrier in Rats. J Med Food. 2020 Nov;23(11):1216-1224. doi: 10.1089/jmf.2019.0247. Epub 2020 Mar 9. PMID 32155356
- [Background] Roldan NR, Jimenez M, Cervantes-Garcia D, Marin E, Salinas E. Glycomacropeptide administration attenuates airway inflammation and remodeling associated to allergic asthma in rat. Inflamm Res. 2016 Apr;65(4):273-83. doi: 10.1007/s00011-015-0913-y. Epub 2016 Jan 11. PMID 26755379
- [Background] Reyes-Pavon D, Cervantes-Garcia D, Bermudez-Humaran LG, Cordova-Davalos LE, Quintanar-Stephano A, Jimenez M, Salinas E. Protective Effect of Glycomacropeptide on Food Allergy with Gastrointestinal Manifestations in a Rat Model through Down-Regulation of Type 2 Immune Response. Nutrients. 2020 Sep 25;12(10):2942. doi: 10.3390/nu12102942. PMID 32992996
- [Background] Munoz FC, Cervantes MM, Cervantes-Garcia D, Jimenez M, Ventura-Juarez J, Salinas E. Glycomacropeptide Attenuates Inflammation, Pruritus, and Th2 Response Associated with Atopic Dermatitis Induced by 2,4-Dinitrochlorobenzene in Rat. J Immunol Res. 2017;2017:6935402. doi: 10.1155/2017/6935402. Epub 2017 Feb 7. PMID 28265582
- [Background] Jimenez M, Chavez NA, Salinas E. Pretreatment with glycomacropeptide reduces allergen sensitization, alleviates immediate cutaneous hypersensitivity and protects from anaphylaxis. Clin Exp Immunol. 2012 Oct;170(1):18-27. doi: 10.1111/j.1365-2249.2012.04631.x. PMID 22943197
- [Background] Wernlund PG, Hvas CL, Dahlerup JF, Bahl MI, Licht TR, Knudsen KEB, Agnholt JS. Casein glycomacropeptide is well tolerated in healthy adults and changes neither high-sensitive C-reactive protein, gut microbiota nor faecal butyrate: a restricted randomised trial. Br J Nutr. 2021 Jun 28;125(12):1374-1385. doi: 10.1017/S0007114520003736. Epub 2020 Sep 24. PMID 32967742
- [Background] Hvas CL, Dige A, Bendix M, Wernlund PG, Christensen LA, Dahlerup JF, Agnholt J. Casein glycomacropeptide for active distal ulcerative colitis: a randomized pilot study. Eur J Clin Invest. 2016 Jun;46(6):555-63. doi: 10.1111/eci.12634. PMID 27090817
- [Background] Ney DM, Etzel MR. Designing medical foods for inherited metabolic disorders: why intact protein is superior to amino acids. Curr Opin Biotechnol. 2017 Apr;44:39-45. doi: 10.1016/j.copbio.2016.10.009. Epub 2016 Nov 16. PMID 27835797
- [Background] Saito T, Itoh T. Variations and distributions of O-glycosidically linked sugar chains in bovine kappa-casein. J Dairy Sci. 1992 Jul;75(7):1768-74. doi: 10.3168/jds.S0022-0302(92)77936-3. PMID 1500573
- [Background] Manthripragada AD, Pinheiro SP, MaCurdy TE, Saneinejad S, Worrall CM, Kelman JA, Graham DJ. Off-label topical calcineurin inhibitor use in children. Pediatrics. 2013 Nov;132(5):e1327-32. doi: 10.1542/peds.2013-0931. Epub 2013 Oct 14. PMID 24127469
- [Background] Ogonowska P, Gilaberte Y, Baranska-Rybak W, Nakonieczna J. Colonization With Staphylococcus aureus in Atopic Dermatitis Patients: Attempts to Reveal the Unknown. Front Microbiol. 2021 Jan 11;11:567090. doi: 10.3389/fmicb.2020.567090. eCollection 2020. PMID 33505363
- [Background] Di Domenico EG, Cavallo I, Bordignon V, Prignano G, Sperduti I, Gurtner A, Trento E, Toma L, Pimpinelli F, Capitanio B, Ensoli F. Inflammatory cytokines and biofilm production sustain Staphylococcus aureus outgrowth and persistence: a pivotal interplay in the pathogenesis of Atopic Dermatitis. Sci Rep. 2018 Jun 28;8(1):9573. doi: 10.1038/s41598-018-27421-1. PMID 29955077
- [Background] Gallegos-Alcala P, Jimenez M, Cervantes-Garcia D, Salinas E. The Keratinocyte as a Crucial Cell in the Predisposition, Onset, Progression, Therapy and Study of the Atopic Dermatitis. Int J Mol Sci. 2021 Oct 1;22(19):10661. doi: 10.3390/ijms221910661. PMID 34639001
- [Background] Al-Khenaizan S. Practical tip: Precooling topical calcineurin inhibitors tube; reduces burning sensation. Dermatol Online J. 2010 Apr 15;16(4):16. PMID 20409423
- [Background] Egeberg A, Schwarz P, Harslof T, Andersen YMF, Pottegard A, Hallas J, Thyssen JP. Association of Potent and Very Potent Topical Corticosteroids and the Risk of Osteoporosis and Major Osteoporotic Fractures. JAMA Dermatol. 2021 Mar 1;157(3):275-282. doi: 10.1001/jamadermatol.2020.4968. PMID 33471030
- [Background] 1. Arenas R. Dermatología, atlas, diagnóstico y tratamiento. 7ma ed. México, Ciudad de México: Mc Graw Hill; 2019.